CLINICAL TRIAL: NCT02107703
Title: MONARCH 2: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of Fulvestrant With or Without Abemaciclib, a CDK4/6 Inhibitor, for Women With Hormone Receptor Positive, HER2 Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) Combined With Fulvestrant in Women With Hormone Receptor Positive HER2 Negative Breast Cancer
Acronym: MONARCH 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15362; I3Y-MC-JPBL (Other: Eli Lilly and Company); 2013-004728-13 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms
Keywords: MONARCH 2
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abemaciclib + Fulvestrant (Experimental): Abemaciclib 150 milligram (mg) administered orally every 12 hours on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500mg administered intramuscularly (IM) on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation were met.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant
- Placebo + Fulvestrant (Placebo Comparator): Placebo administered orally every 12 hours on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500mg administered IM on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation were met.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Administered Orally
  Other Names: LY2835219
  Arms: Abemaciclib + Fulvestrant
Drug: Fulvestrant — Administered IM
Drug: Placebo — Administered Orally
  Arms: Placebo + Fulvestrant

SUMMARY:
The main purpose of this study is to compare progression-free survival for women with hormone receptor positive (HR+), human epidermal growth factor receptor (HER2) negative advanced breast cancer receiving either abemaciclib + fulvestrant or fulvestrant alone. Participants will be randomized to abemaciclib or placebo in a 2:1 ratio. The study will last about 9 months for each participant.

For the endocrine naïve cohort, all participants will received abemaciclib + fulvestrant.

ELIGIBILITY:
Inclusion Criteria

* Have a diagnosis of HR+, HER2- breast cancer
* Have locally advanced disease not amenable to curative treatment by surgery or metastatic disease. In addition, participants must fulfill 1 of the following criteria:

  * relapsed with radiologic evidence of progression while receiving neoadjuvant or adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression
  * relapsed with radiologic evidence of progression within 1 year from completion of adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression
  * relapsed with radiologic evidence of progression more than 1 year from completion of adjuvant endocrine therapy and then subsequently relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease. Participants may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease
  * presented de novo with metastatic disease and then relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as first line endocrine therapy for metastatic disease. Participants may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease
  * for the endocrine naïve cohort: Must not have received prior endocrine therapy in current or prior disease setting
* Have postmenopausal status due to either surgical/natural menopause or ovarian suppression (initiated at least 28 days prior to Day 1 of Cycle 1) with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin
* Have a negative serum pregnancy test at baseline (within 14 days prior to randomization) and agree to use medically approved precautions to prevent pregnancy during the study and for 12 weeks following the last dose of abemaciclib if postmenopausal status is due to ovarian suppression with a GnRH agonist
* Have either measurable disease or nonmeasurable bone only disease
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued previous therapies for cancer (including specifically, aromatase inhibitors, anti-estrogens, chemotherapy, radiotherapy, and immunotherapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (until the toxicity resolves to either baseline or at least Grade 1) except for residual alopecia or peripheral neuropathy

Exclusion Criteria

* Are currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis visceral crisis is not the mere presence of visceral metastases but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of the disease
* Have clinical evidence or history of central nervous system metastasis
* Have received prior treatment with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy), fulvestrant, everolimus, or any CDK4/6 inhibitor. For the endocrine naïve cohort: In addition, have received treatment with any prior endocrine therapy
* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days prior to randomization of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively
* Have received recent (within 28 days prior to randomization) yellow fever vaccination
* Have had major surgery within 14 days prior to randomization of study drug to allow for post-operative healing of the surgical wound and site(s)
* Have a personal history within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest
* Have inflammatory breast cancer or a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years
* Have received an autologous or allogeneic stem-cell transplant
* Have active bacterial or fungal infection, or detectable viral infection
* Have initiated bisphosphonates or approved Receptor activator of nuclear factor kappa-B (RANK) ligand targeted agents <7 days prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (144):
- United States (41):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - University of California - San Diego, La Jolla, California
  - Kaiser Permanente, Riverside, California
  - Univ of California San Francisco, San Francisco, California
  - Stanford University Clinic, Stanford, California
  - Palm Beach Cancer Institue, Atlantis, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Palm Beach Cancer Institue, Palm Beach Gardens, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center, Tampa, Florida
  - Palm Beach Cancer Institue, Wellington, Florida
  - Palm Beach Cancer Institue, West Palm Beach, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Harbin Clinic, Rome, Georgia
  - Quincy Medical Group, Quincy, Illinois
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Breslin Cancer Center, Lansing, Michigan
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - Washington University Medical School, City of Saint Peters, Missouri
  - Washington University Medical School, Creve Coeur, Missouri
  - Freeman Cancer Institute, Joplin, Missouri
  - St Lukes Hospital, Kansas City, Missouri
  - Washington University Medical School, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Novant Health, Oncology Research Institute, Winston-Salem, North Carolina
  - Oklahoma Cancer Specialists & Research Institute, LLC, Tulsa, Oklahoma
  - Sanford Research/USD, Sioux Falls, South Dakota
  - The Boston Baskin Cancer Group, Memphis, Tennessee
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - St Mary Regional Cancer Center, Walla Walla, Washington
- Australia (5):
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Monash Cancer Centre, East Bentleigh, Victoria
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (4):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Canada (4):
  - Tom Baker Cancer Center, Calgary, Alberta
  - London Regional Cancer Program, London, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
- Denmark (3):
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Aalborg Universitets hospital, Aalborg
  - Roskilde Sygehus, Roskilde
- Finland (3):
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Uusimaa
  - Turun Yliopistollinen Keskussairaala, Turku
- France (4):
  - CHU Besançon, Besançon, Doubs
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand, Puy-de-Dôme
  - Polyclinique De Blois, La Chaussée-Saint-Victor
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
- Germany (5):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Gemeinschaftspraxis hop-augsburg, Augsburg, Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Facharztzentrum Eppendorf, Hamburg
- Greece (4):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Krítí
  - Chania General Hospital 'Agios Georgios', Chania
- Italy (4):
  - Azienda Ospedaliero Universitaria S.Anna, Cona, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Ospedale Bellaria - Azienda USL di Bologna, Bologna
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (19):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume General Hospital, Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Met Cancer & Infectious Diseases Center Komagome Hp, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Sagara Hospital, Kagoshima
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Osaka Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (7):
  - Hospital Angeles, Tijuana, Estado de Baja California
  - Preparaciones Oncológicas S.C., León, Guanajuato
  - Centro Oncológico Internacional (COI), Guadalajara, Jalisco
  - Grupo Medico Camino Sc, Mexico City, Mexico City
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - OCA Hospital, Monterrey, Nuevo León
  - Tecnologico de Monterrey, Monterrey, Nuevo León
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Bialostockie Centrum Onkologii, Oddzial Onkologii Klinicznej, Bialystok
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Puerto Rico Hematology/Oncology Group, Bayamón, PR, Puerto Rico
- Romania (3):
  - S.C. MedisProf SRL, Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Ianuli Med Consult SRL, Bucharest
- Russia (6):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Regional Budgetary Healthcare Institution 'Ivanovo Regional Oncology Dispensary', Ivanovo, Ivanovo Oblast
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moscow, Moscow
  - Kursk Regional Oncology Dispensary, Kursk, Russian Federation
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg, Sankt-Peterburg
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (7):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [Lérida]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia, Región de
  - Hospital Quirónsalud Valencia, Valencia, València
  - Hospital Clinico San Carlos, Madrid
- Switzerland (3):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Spital Thun, Thun, Canton of Bern
  - HUG-Hôpitaux Universitaires de Genève, Geneva
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Neven P, Rugo HS, Tolaney SM, Iwata H, Toi M, Goetz MP, Kaufman PA, Lu Y, Haddad N, Hurt KC, Sledge GW Jr. Abemaciclib plus fulvestrant in hormone receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer in premenopausal women: subgroup analysis from the MONARCH 2 trial. Breast Cancer Res. 2021 Aug 23;23(1):87. doi: 10.1186/s13058-021-01463-2. PMID 34425869
- [Derived] Inoue K, Masuda N, Iwata H, Takahashi M, Ito Y, Miyoshi Y, Nakayama T, Mukai H, van der Walt JS, Mori J, Sakaguchi S, Kawaguchi T, Tanizawa Y, Llombart-Cussac A, Sledge GW Jr, Toi M. Japanese subpopulation analysis of MONARCH 2: phase 3 study of abemaciclib plus fulvestrant for treatment of hormone receptor-positive, human epidermal growth factor receptor 2-negative breast cancer that progressed on endocrine therapy. Breast Cancer. 2021 Sep;28(5):1038-1050. doi: 10.1007/s12282-021-01239-8. Epub 2021 Apr 1. PMID 33797023
- [Derived] Goetz MP, Okera M, Wildiers H, Campone M, Grischke EM, Manso L, Andre VAM, Chouaki N, San Antonio B, Toi M, Sledge GW Jr. Safety and efficacy of abemaciclib plus endocrine therapy in older patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: an age-specific subgroup analysis of MONARCH 2 and 3 trials. Breast Cancer Res Treat. 2021 Apr;186(2):417-428. doi: 10.1007/s10549-020-06029-y. Epub 2021 Jan 3. PMID 33392835
- [Derived] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Conte P, Lu Y, Barriga S, Hurt K, Frenzel M, Johnston S, Llombart-Cussac A. The Effect of Abemaciclib Plus Fulvestrant on Overall Survival in Hormone Receptor-Positive, ERBB2-Negative Breast Cancer That Progressed on Endocrine Therapy-MONARCH 2: A Randomized Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):116-124. doi: 10.1001/jamaoncol.2019.4782. PMID 31563959
- [Derived] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Frenzel M, Lin Y, Barriga S, Smith IC, Bourayou N, Llombart-Cussac A. MONARCH 2: Abemaciclib in Combination With Fulvestrant in Women With HR+/HER2- Advanced Breast Cancer Who Had Progressed While Receiving Endocrine Therapy. J Clin Oncol. 2017 Sep 1;35(25):2875-2884. doi: 10.1200/JCO.2017.73.7585. Epub 2017 Jun 3. PMID 28580882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: With Overall Survival (OS) as a key outcome, participants who completed included those who died due to any cause and those who were off treatment, alive and in follow-up at the time of the final OS analysis.
Period: Overall Study
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Started | 446 | 223
Received at Least 1 Dose of Study Drug | 441 | 223
Completed | 332 | 188
Not Completed | 114 | 35
Not completed — Withdrawal by Subject | 46 | 21
Not completed — Lost to Follow-up | 20 | 9
Not completed — On study treatment/follow up | 48 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Abemaciclib + Fulvestrant: Abemaciclib 150 mg administered orally every 12 hours on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500mg administered intramuscularly (IM) on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation were met.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 446 | 223 | 669
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.2) | 61.1 (11.7) | 59.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 446 | 223 | 669
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants who had baseline Ethnicity data.
  Participants
    number analyzed (Participants) | 443 | 223 | 666
    Hispanic or Latino | 57 | 25 | 82
    Not Hispanic or Latino | 303 | 162 | 465
    Unknown or Not Reported | 83 | 36 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 8 | 26
  Asian | 149 | 65 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 237 | 136 | 373
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 9 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 120 | 58 | 178
  Europe | 179 | 100 | 279
  Taiwan | 25 | 14 | 39
  Japan | 64 | 31 | 95
  South Korea | 58 | 20 | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: From Date of Randomization until Disease Progression or Death Due to Any Cause (Up To 31 Months)
Population: All randomized participants. Censored participants: Abemaciclib=224.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Abemaciclib + Fulvestrant: Abemaciclib 150 mg administered orally every 12 hours on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500mg administered IM on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation were met.
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 446 | 223
Months | 16.4 [14.4 to 19.3] | 9.3 [7.4 to 11.4]
Statistical Analysis 1: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; The final analysis was planned at 378 PFS events, which would provide approximately 90% power assuming a hazard ratio (HR) of 0.703 at a one-sided α of 0.025; Test type: Other; p < 0.0000001, Log Rank — This is two sided P value and it is statistically significant; Log rank test is stratified by endocrine sensitivity and natural of disease by interactive web response system (IWRS); Hazard Ratio (HR) = 0.553, 95% CI 2-sided [0.449 to 0.681]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of randomization to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive. The final analysis of the OS outcome was conducted after 440 OS events had been observed.
Time Frame: From Date of Randomization until Death Due to Any Cause (Up To 72 Months)
Population: All randomized participants. Censored participants: Abemaciclib=163 (36.5%), Placebo = 66 (29.6).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 446 | 223
Months | 45.80 [38.96 to 52.64] | 37.25 [34.36 to 43.20]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 31 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 446 | 223
Percentage of participants | 35.2 [30.8 to 39.6] | 16.1 [11.3 to 21.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of CR, PR until Disease Progression or Death Due to Any Cause (Up To 31 Months)
Population: All randomized participants with response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 157 | 36
Months | NA [18.05 to NA] — The median DoR for participants has not been reached. | 25.6 [11.9 to 25.6]

5. Secondary Outcome: Percentage of Participants Achieving CR, PR or Stable Disease (SD) (Disease Control Rate [DCR])
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 31 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 446 | 223
Percentage of participants | 83.0 [79.5 to 86.4] | 75.8 [70.2 to 81.4]

6. Secondary Outcome: Percentage of Participants With CR, PR or SD With a Duration of At Least 6 Months (Clinical Benefit Rate [CBR])
Description: Clinical benefit rate defined as percentage of participants with best overall response of CR, PR, or SD with a duration of at least 6 months.CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions.PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Percentage of participants=(participants with CR+PR+SD with a duration of at least 6 months /number of participants enrolled) *100.PD was at least a 20% increase in sum of the diameters of target lesions,with reference being the smallest sum on study and an absolute increase of at least 5 mm or unequivocal progression of non-target lesions,or 1 or more new lesions.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 31 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 446 | 223
Percentage of participants | 72.2 [68.0 to 76.4] | 56.1 [49.5 to 62.6]

7. Secondary Outcome: Change From Baseline in Pain and Symptom Burden Assessment Using the Modified Brief Pain Inventory-Short Form (mBPI-sf)
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). The overall change is based on the estimated main treatment effect. Least square (LS) Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, End of Study (Up To 31 Months)
Population: All randomized participants who received at least one dose of study drug with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 441 | 223
score on a scale | -0.06 (0.07) | 0.00 (0.10)

8. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of Abemaciclib, Its Metabolites M2 and M20
Description: Area Under the Plasma Concentration versus Time Curve from Time Zero to Infinity (AUC[0-∞]) was evaluated for Abemaciclib and Metabolites M2 and M20.
Time Frame: Cycle 1 Day 1 2-4 hours (h) post dose, Cycle 1 Day 15 4 and 7h post dose, Cycle 2 Day 1 pre dose and 3h post dose, Cycle 3 Day1 pre dose
Population: All randomized participants who received at least one dose of 150 mg study drug (Abemaciclib) with evaluable Abemaciclib, M2 and M20 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour/milliliters (ng*h/mL)
Arm/Group | Abemaciclib + Fulvestrant
Number analyzed (Participants) | 326
Nanograms*hour/milliliters (ng*h/mL)
  Abemaciclib | 2960 (32.2)
  M2 | 1640 (70.2)
  M20 | 2870 (69.6)

9. Secondary Outcome: Change From Baseline in Health Status Using the EuroQol 5-Dimension 5 Level (EQ-5D 5L)
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The EQ-5D-5L is assessed using a visual analog scale (VAS) that ranged from 0 to 100mm, where 0 is the worst health you can imagine and 100 is the best health you can imagine. A higher score indicates better health state. LS Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, End of Study (Up To 31 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 5L data.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 441 | 223
mm | 0.12 (0.65) | 1.16 (0.92)

10. Secondary Outcome: Change From Baseline to Short Term Follow up in Quality of Life Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, scores range from 0 to 110 with higher scores representing a better level of functioning. For symptoms scales, scores range from 0 to 100 with higher scores representing a greater degree of symptoms. LS Mean value of changing from baseline to short follow up was estimated from the mixed model that was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, Short Term Follow Up (Up To 31 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-C30 data at short term follow up for each EORTC QLQ-C30 items.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 180 | 126
units on a scale
  Global health status: number analyzed (Participants) | 179 | 126
  Global health status | -4.57 (1.55) | -8.15 (1.87)
  Functional scale: Physical functioning: number analyzed (Participants) | 179 | 126
  Functional scale: Physical functioning | -3.76 (1.29) | -7.59 (1.59)
  Functional scale: Role functioning: number analyzed (Participants) | 179 | 124
  Functional scale: Role functioning | -4.87 (1.73) | -9.58 (2.12)
  Functional scale: Emotional functioning: number analyzed (Participants) | 179 | 125
  Functional scale: Emotional functioning | 2.38 (1.38) | -2.44 (1.70)
  Functional scale: Cognitive functioning: number analyzed (Participants) | 180 | 125
  Functional scale: Cognitive functioning | -3.16 (1.29) | -2.96 (1.58)
  Functional scale: Social functioning | -4.62 (1.61) | -4.78 (1.97)
  Symptom scale: Fatigue: number analyzed (Participants) | 180 | 125
  Symptom scale: Fatigue | 5.01 (1.45) | 7.83 (1.78)
  Symptom scale: Nausea and vomiting: number analyzed (Participants) | 180 | 125
  Symptom scale: Nausea and vomiting | 2.81 (1.35) | 6.49 (1.64)
  Symptom scale: Pain | -0.47 (1.82) | 4.38 (2.21)
  Symptom scale: Dyspnoea: number analyzed (Participants) | 180 | 123
  Symptom scale: Dyspnoea | 5.21 (1.70) | 5.39 (2.10)
  Symptom scale: Insomnia | -0.04 (1.86) | 3.76 (2.27)
  Symptom scale: Appetite loss: number analyzed (Participants) | 180 | 125
  Symptom scale: Appetite loss | 2.06 (1.85) | 6.40 (2.23)
  Symptom scale: Constipation: number analyzed (Participants) | 179 | 125
  Symptom scale: Constipation | -0.15 (1.59) | 3.79 (1.92)
  Symptom scale: Diarrhoea: number analyzed (Participants) | 179 | 125
  Symptom scale: Diarrhoea | 4.14 (1.66) | 2.67 (1.99)
  Symptom scale: Financial difficulties: number analyzed (Participants) | 179 | 124
  Symptom scale: Financial difficulties | 0.34 (1.60) | 2.85 (1.96)

11. Secondary Outcome: Change From Baseline to Short Term Follow up in Quality of Life Using the EORTC QLQ-BR23 (Breast) Questionnaire
Description: EORTC-QLQ-BR23 measured multi-item functional scales for body image, sexual functioning and future perspective and measured single item symptoms scales which assessed systemic therapy side effects, breast symptoms and arm symptoms. For functional scales, scores ranged from 0 to 100 where higher scores represented a better level of functioning. For symptoms scales, scores ranged from 0 to 100 where higher scores represented a greater degree of symptoms. LS Mean value of changing from baseline to short follow up was estimated from the mixed model that was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, Short Term Follow Up (Up To 31 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-BR23 data at short term follow up for each BR23 items.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 182 | 126
Units on a scale
  Functional scale: Body image: number analyzed (Participants) | 179 | 125
  Functional scale: Body image | -2.20 (1.46) | -3.27 (1.83)
  Functional scale:Sexual functioning: number analyzed (Participants) | 171 | 116
  Functional scale:Sexual functioning | 0.41 (1.00) | -1.60 (1.25)
  Functional scale: Future perspective: number analyzed (Participants) | 179 | 126
  Functional scale: Future perspective | 6.06 (2.06) | 10.05 (2.51)
  Symptom scale: Systemic therapy side effects: number analyzed (Participants) | 182 | 125
  Symptom scale: Systemic therapy side effects | 7.23 (1.00) | 6.98 (1.22)
  Symptom scale: Breast symptoms: number analyzed (Participants) | 181 | 126
  Symptom scale: Breast symptoms | -2.10 (0.89) | -0.96 (1.09)
  Symptom scale: Arm symptoms: number analyzed (Participants) | 182 | 125
  Symptom scale: Arm symptoms | -0.45 (1.29) | 0.10 (1.59)

ADVERSE EVENTS:
Time Frame: Up To 7 years 7.7 Months
Description: Adverse Events: All randomized participants who received at least one dose of study drug; All-Cause Mortality: All randomized participants. Analyses presented in this report are based on a database lock for the pre-planned final OS analysis of 22 April 2022.
Groups:
- Abemaciclib + Fulvestrant: 150 mg Abemaciclib given orally once every 12 hours in 28 day cycles. 500 mg fulvestrant administered as two 250-mg injections intramuscularly (IM) on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 283/446 | 157/223
Serious Adverse Events (participants affected / at risk) | 129/441 | 33/223
Other Adverse Events (participants affected / at risk) | 432/441 | 194/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Fulvestrant (N=441) | Placebo + Fulvestrant (N=223)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (13) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 1 (1)
Skin infection (Infections and infestations) | 6 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 0 (0)
Blood follicle stimulating hormone abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Hormone level abnormal (Investigations) | 1 (1) | 0 (0)
Oestradiol abnormal (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 9 (11) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Fulvestrant (N=441) | Placebo + Fulvestrant (N=223)
Anaemia (Blood and lymphatic system disorders) | 155 (313) | 11 (15)
Leukopenia (Blood and lymphatic system disorders) | 148 (500) | 4 (10)
Lymphopenia (Blood and lymphatic system disorders) | 45 (113) | 2 (9)
Neutropenia (Blood and lymphatic system disorders) | 219 (760) | 8 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 79 (135) | 6 (7)
Lacrimation increased (Eye disorders) | 34 (44) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 24 (28) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 166 (320) | 36 (65)
Constipation (Gastrointestinal disorders) | 73 (96) | 36 (47)
Diarrhoea (Gastrointestinal disorders) | 384 (1205) | 62 (104)
Dry mouth (Gastrointestinal disorders) | 35 (40) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 33 (43) | 12 (15)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 (27) | 5 (5)
Nausea (Gastrointestinal disorders) | 218 (367) | 55 (72)
Stomatitis (Gastrointestinal disorders) | 82 (119) | 24 (30)
Vomiting (Gastrointestinal disorders) | 130 (253) | 26 (43)
Chills (General disorders) | 26 (30) | 1 (1)
Fatigue (General disorders) | 192 (294) | 64 (81)
Influenza like illness (General disorders) | 41 (71) | 16 (23)
Injection site reaction (General disorders) | 48 (66) | 22 (40)
Oedema peripheral (General disorders) | 62 (83) | 16 (21)
Pain (General disorders) | 30 (42) | 11 (14)
Pyrexia (General disorders) | 62 (99) | 16 (18)
Sinusitis (Infections and infestations) | 24 (36) | 6 (7)
Skin infection (Infections and infestations) | 25 (36) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 88 (159) | 19 (32)
Urinary tract infection (Infections and infestations) | 46 (76) | 10 (18)
Alanine aminotransferase increased (Investigations) | 79 (138) | 12 (15)
Aspartate aminotransferase increased (Investigations) | 81 (132) | 16 (25)
Blood alkaline phosphatase increased (Investigations) | 27 (47) | 7 (10)
Blood creatinine increased (Investigations) | 63 (134) | 1 (1)
Weight decreased (Investigations) | 54 (65) | 7 (10)
Decreased appetite (Metabolism and nutrition disorders) | 127 (162) | 30 (31)
Hypokalaemia (Metabolism and nutrition disorders) | 41 (77) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 (154) | 34 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 62 (100) | 30 (40)
Bone pain (Musculoskeletal and connective tissue disorders) | 29 (36) | 21 (25)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 53 (90) | 15 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 44 (57) | 14 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 (119) | 11 (13)
Dizziness (Nervous system disorders) | 67 (111) | 16 (18)
Dysgeusia (Nervous system disorders) | 82 (106) | 6 (7)
Headache (Nervous system disorders) | 108 (203) | 36 (67)
Neuropathy (Nervous system disorders) | 42 (51) | 21 (26)
Anxiety (Psychiatric disorders) | 23 (26) | 5 (6)
Depression (Psychiatric disorders) | 26 (28) | 10 (12)
Insomnia (Psychiatric disorders) | 42 (53) | 21 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 78 (114) | 30 (35)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 (58) | 23 (28)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (32) | 14 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 76 (88) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 23 (29) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 48 (61) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 64 (82) | 16 (18)
Rash (Skin and subcutaneous tissue disorders) | 54 (75) | 11 (13)
Embolism (Vascular disorders) | 26 (31) | 1 (1)
Hot flush (Vascular disorders) | 51 (71) | 25 (28)
Lymphoedema (Vascular disorders) | 23 (25) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (8):
  • Study Protocol: JPBL 05 Protocol_Redacted (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_000.pdf
  • Study Protocol: JPBL 05 Protocol (a)_Redacted (2015-01-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_001.pdf
  • Study Protocol: JPBL 05 Protocol (b)_Redacted (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_002.pdf
  • Study Protocol: JPBL 05 Protocol (c)_Redacted (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_003.pdf
  • Study Protocol: JPBL 05 Protocol (d)_Redacted (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_004.pdf
  • Study Protocol: JPBL 05 Protocol (g)_Redacted (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/Prot_007.pdf
  • Statistical Analysis Plan: version 4 (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/SAP_005.pdf
  • Statistical Analysis Plan: Addendum for Overall Survival Analyses (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02107703/SAP_006.pdf